CLINICAL TRIAL: NCT03761316
Title: Goal Setting in SCS Patients: a Qualitative Review (LEISURE)
Brief Title: Goal Setting in SCS Patients: a Qualitative Review
Status: Completed | Type: Observational
Sponsor: Moens Maarten (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Moens Maarten, Prof. dr., Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Other Study IDs: LEISURE
Record Dates: First submitted 2018-11-28; First posted 2018-12-03 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Failed Back Surgery Syndrome
Keywords: Spinal cord stimulation; interview
MeSH Terms: conditions — Failed Back Surgery Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FBSS patients: patients with Failed Back Surgery Syndrome, eligible for SCS
  Interventions: Other: interview regarding goals

INTERVENTIONS:
Other: interview regarding goals — interview regarding goals

SUMMARY:
This is a prospective study in which the investigators will describe individual goals of patients with Failed Back Surgery Syndrome, who will be treated with spinal cord stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain as a result of FBSS that exists for at least 6 months with a pain intensity 5 or higher measured on numeric rating scale (NRS)
* FBSS patients suitable for SCS
* Age > 18 years
* Native Dutch or French speeking patients

Exclusion Criteria:

* Expected inability of patients to receive or properly operate the spinal cord stimulation system
* History of coagulation disorders, lupus erythematosus, diabetic neuropathy, rheumatoid arthritis or morbus Bechterew
* Active malignancy
* Addiction to any of the following drugs, alcohol (5E/day) and/or medication
* Evidence of an active disruptive psychiatric disorder or other known condition significant enough to impact perception of pain, compliance to intervention and/or ability to evaluate treatment outcome as determined by investigator
* Immune deficiency (HIV positive, immunosuppressiva, etc.)
* Life expectancy < 1 year
* Local infection or other skin disorder at site of incision
* Pregnancy
* Other implanted active medical device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with medication-resistant chronic back and leg pain due to Failed Back Surgery Syndrome who are offered treatment with SCS.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Goals and expectations towards spinal cord stimulation | Before spinal cord stimulation implantation
  Individual goals and expectations regarding the treatment with spinal cord stimulation will be explored during an interview

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Moens, Prof. dr., Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium